CLINICAL TRIAL: NCT04660318
Title: Assessment of Physiological Parameters Measurements (Heart Rate, Respiratory Rate, and Oxygen Saturation) by Standard Acquisition System Compared Remote Photoplethysmography Imaging System
Brief Title: Assessment of Physiological Parameters Measurements (Heart Rate, Respiratory Rate, and Oxygen Saturation) by Standard Acquisition System Compared Remote Photoplethysmography Imaging System l
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02428-31
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Plethysmography; Remote Photoplethysmography Imaging; Physiological Parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: remote photoplethysmography for physiological parameters Monitor Readings (Experimental)
  Interventions: Device: Remote photoplethysmography for physiological parameters
- Control: rstandard acquisition system for physiological parameters Monitor Readings (Other)
  Interventions: Device: standard acquisition system for physiological parameters

INTERVENTIONS:
Device: Remote photoplethysmography for physiological parameters — physiological parameters will be acquired using the Remote photoplethysmography software simultaneously for the conventional parameters measurements (heart rate, respiratory rate, and oxygen saturation)
  Arms: Experimental: remote photoplethysmography for physiological parameters Monitor Readings
Device: standard acquisition system for physiological parameters — physiological parameters will be acquired using the standard acquisition system for the conventional parameters measurements (heart rate, respiratory rate, and oxygen saturation)
  Arms: Control: rstandard acquisition system for physiological parameters Monitor Readings

SUMMARY:
Introduced in 1930, photoplethysmography techniques presented the possibility of measuring SpO2 and HR using the absorption of light by the blood to define these signals In recent years, a new approach to photoplethysmography to measure physiological parameters without contact has been developed. This technique, called remote Photoplethysmography Imaging (rPPG), uses the different Red - Green - Blue color spectra at a skin captured by the camera video to determine a plethysmography signal.

Although these systems have been technically valid, they have not been clinically evaluated in a health setting. This clinical trial is to assess parameters measurements by rPPG compared standard acquisition system in real conditions

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a Pulmonary function testing.

Exclusion Criteria:

* Patients with stable clinical status.
* Pregnant woman or Woman of childbearing potential without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1045 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Concordance of rPPG heart rate readings | 30-120 seconds.
  Heart rateconcordance analysis by standard acquisition system (photoplethysmography of the finger) compared rPPG
Concordance of rPPG respiratory rate readings | 30-120 seconds.
  respiratory rate concordance analysis by standard acquisition system (photoplethysmography of the finger) compared rPPG
Concordance of rPPG oxygen saturation readings | 30-120 seconds.
  oxygen saturation concordance analysis by standard acquisition system (photoplethysmography of the finger) compared rPPG

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy., Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Allado E, Poussel M, Moussu A, Saunier V, Bernard Y, Albuisson E, Chenuel B. Innovative measurement of routine physiological variables (heart rate, respiratory rate and oxygen saturation) using a remote photoplethysmography imaging system: a prospective comparative trial protocol. BMJ Open. 2021 Aug 13;11(8):e047896. doi: 10.1136/bmjopen-2020-047896. PMID 34389569